CLINICAL TRIAL: NCT00474968
Title: Clinical Study Validating the Adequacy, Efficacy, and Safety of the e2TM Cervical Cell Collector Compared to Standard Spatula/CytoBrush Technique In Patients With Recent History of Abnormal Pap Test Returning for Colposcopy/Biopsy.
Brief Title: Adequacy and Efficacy of the e2TM Cervical Cell Collector Compared to Standard Spatula/CytoBrush Technique.
Status: Completed | Type: Observational
Sponsor: CytoCore, Inc. (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Richard Domanik, CytoCore
Other Study IDs: e2TM Cervical cell Collector
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Colposcopy; Biopsy
MeSH Terms: interventions — Toothbrushing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Cervical cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arm 1 - Experimental: e2 Cell Collector [SoftPAP(R)]
  Interventions: Device: e2 Cell Collector [SoftPAP(R)]
- Arm 2 - Control: Brush/spatula
  Interventions: Device: Spatula/Brush

INTERVENTIONS:
Device: e2 Cell Collector [SoftPAP(R)] — Cervical cells collected using the e2 Cell Collector [SoftPAP(R)]
  Groups: Arm 1 - Experimental
Device: Spatula/Brush — Cervical cells collected using a combination of a cervical spatula and an endocervical brush
  Groups: Arm 2 - Control

SUMMARY:
A clinical study to determine the adequacy and efficacy of the InPath e2TM Collector compared to the FDA-approved spatula/cytobrush when used as the cell collection device in screening for cervical cancer.

The InPath e2TM Collector name has been changed to the CytoCore SoftPAP(R) Collector

DETAILED DESCRIPTION:
The e2TM (SoftPAP) Collector collects only cells that have been exfoliated from the cervix whereas spatulas, brushes and broom-style collection devices collect cells by scraping or abrading the cervix. THis trial is to determine whether the purely exfoliated sample collected using the e2TM Collector is equivalent to samples obtained by scraping or abrading the cervix for purposes of cervical cancer screening and HPV detection.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 years old and above
* Women scheduled to undergo colposcopy

Exclusion Criteria:

* Patients who have had a hysterectomy
* Patients who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women > 18 years of age with an abnormal pap within 30 days to 1 year for whom a colposcopy is scheduled.
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay S. Pinkerton, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (7):
- United States (7):
  - Visions Clinical Research, Wellington, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - St. Louis University, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh Medical Centers, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Fort Worth, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Sankaranarayanan R, Budukh AM, Rajkumar R. Effective screening programmes for cervical cancer in low- and middle-income developing countries. Bull World Health Organ. 2001;79(10):954-62. Epub 2001 Nov 1. PMID 11693978
- [Background] Waxman AG. Guidelines for cervical cancer screening: history and scientific rationale. Clin Obstet Gynecol. 2005 Mar;48(1):77-97. doi: 10.1097/01.grf.0000151590.08451.26. No abstract available. PMID 15725861
- [Background] Holowaty P, Miller AB, Rohan T, To T. RESPONSE: re: natural history of dysplasia of the uterine cervix. J Natl Cancer Inst. 1999 Aug 18;91(16):1420A-1421. doi: 10.1093/jnci/91.16.1420a. No abstract available. PMID 10451450
- [Background] Solomon D, Davey D, Kurman R, Moriarty A, O'Connor D, Prey M, Raab S, Sherman M, Wilbur D, Wright T Jr, Young N; Forum Group Members; Bethesda 2001 Workshop. The 2001 Bethesda System: terminology for reporting results of cervical cytology. JAMA. 2002 Apr 24;287(16):2114-9. doi: 10.1001/jama.287.16.2114. PMID 11966386
- [Background] Nanda K, McCrory DC, Myers ER, Bastian LA, Hasselblad V, Hickey JD, Matchar DB. Accuracy of the Papanicolaou test in screening for and follow-up of cervical cytologic abnormalities: a systematic review. Ann Intern Med. 2000 May 16;132(10):810-9. doi: 10.7326/0003-4819-132-10-200005160-00009. PMID 10819705
- [Background] Fahey MT, Irwig L, Macaskill P. Meta-analysis of Pap test accuracy. Am J Epidemiol. 1995 Apr 1;141(7):680-9. doi: 10.1093/oxfordjournals.aje.a117485. PMID 7702044
- [Background] Clavel C, Masure M, Bory JP, Putaud I, Mangeonjean C, Lorenzato M, Nazeyrollas P, Gabriel R, Quereux C, Birembaut P. Human papillomavirus testing in primary screening for the detection of high-grade cervical lesions: a study of 7932 women. Br J Cancer. 2001 Jun 15;84(12):1616-23. doi: 10.1054/bjoc.2001.1845. PMID 11401314
- [Background] Willis BH, Barton P, Pearmain P, Bryan S, Hyde C. Cervical screening programmes: can automation help? Evidence from systematic reviews, an economic analysis and a simulation modelling exercise applied to the UK. Health Technol Assess. 2005 Mar;9(13):1-207, iii. doi: 10.3310/hta9130. PMID 15774236
- [Background] Buntinx F, Brouwers M. Relation between sampling device and detection of abnormality in cervical smears: a meta-analysis of randomised and quasi-randomised studies. BMJ. 1996 Nov 23;313(7068):1285-90. doi: 10.1136/bmj.313.7068.1285. PMID 8942687
- [Background] Martin-Hirsch P, Lilford R, Jarvis G, Kitchener HC. Efficacy of cervical-smear collection devices: a systematic review and meta-analysis. Lancet. 1999 Nov 20;354(9192):1763-70. doi: 10.1016/s0140-6736(99)02353-3. PMID 10577637
- [Background] Martin-Hirsch P, Jarvis G, Kitchener H, Lilford R. Collection devices for obtaining cervical cytology samples. Cochrane Database Syst Rev. 2000;2000(2):CD001036. doi: 10.1002/14651858.CD001036. PMID 10796736
- [Background] Selvaggi SM, Guidos BJ. Specimen adequacy and the ThinPrep Pap Test: the endocervical component. Diagn Cytopathol. 2000 Jul;23(1):23-6. doi: 10.1002/1097-0339(200007)23:13.0.CO;2-K. PMID 10907927
- [Background] Marchand L, Mundt M, Klein G, Agarwal SC. Optimal collection technique and devices for a quality pap smear. WMJ. 2005 Aug;104(6):51-5. PMID 16218317
- [Background] Koss LG. Evolution in cervical pathology and cytology: a historical perspective. Eur J Gynaecol Oncol. 2000;21(6):550-4. No abstract available. PMID 11214608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting for a previously scheduled colposcopy subsequent to an abnormal Pap result were recruited for this study.
Groups:
- SoftPAP: Samples collected using the SoftPAP Collector
- Brush/Spatula: Samples collected using an endocervical brush and cervical spatula
Period: Overall Study
Arm/Group | SoftPAP | Brush/Spatula
Started | 366 | 371
Completed | 348 | 355
Not Completed | 18 | 16
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Protocol Violation | 9 | 8
Not completed — Sample not collected | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SoftPAP | Brush/Spatula | Total
Number analyzed (Participants) | 366 | 371 | 737
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 366 | 365 | 731
  >=65 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366 | 371 | 737
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 366 | 371 | 737

OUTCOME MEASURES:

1. Primary Outcome: Cell Collection Efficacy
Description: True Positive (TP); True Negative (TN), False Positive (FP) and False Negative (FN) participants and percentage of participants based upon comparison of the cytology diagnosis (Dx) with biopsy (Bx) and endocervical curretage (ECC) results from the same patient.
Time Frame: At the time of cell collection.
Population: 79/348 (Arm 1) and 81/355 (Arm 2) participants were excluded from the sensitivity/specificity analysis due to biopsy (Bx) and/or endocervical curettage (ECC) results not being reported
Measure: Number; unit: Participants
Arm/Group | SoftPAP | Brush/Spatula
Number analyzed (Participants) | 348 | 355
Participants
  True Positive (TP) (Cytology Dx vs (Bx + ECC) | 174 | 170
  True Negative (TN) (Cytology Dx vs (Bx + ECC)) | 33 | 14
  False Positive (FP) (Cytology Dx vs (Bx + ECC)) | 42 | 63
  False Negative (FN) (Cytology Dx vs (Bx + ECC)) | 20 | 27
  Excluded - Bx/ECC results not reported | 79 | 81

2. Secondary Outcome: Human Papilloma Virus (HPV) Detection Frequency
Description: Number and percentage of HPV positive specimens by the Hybrid Capture II (HC-II) assay
Time Frame: At the time of cell collection.
Measure: Number; unit: Participants
Arm/Group | SoftPAP | Brush/Spatula
Number analyzed (Participants) | 348 | 355
Participants
  HPV Positive by Hybrid Capture-II | 165 | 214
  HPV Negative by Hybrid Capture-II | 82 | 104
  Hybrid Capture-II Results Not Reported | 101 | 37

3. Primary Outcome: Specimen Adequacy
Description: Number and percentage of samples classified as adequate for diagnosis
Time Frame: At time of cell collection
Population: Includes all cytology specimens
Measure: Number; unit: Participants
Arm/Group | SoftPAP | Brush/Spatula
Number analyzed (Participants) | 348 | 355
Participants
  Satisfactory for Diagnosis | 343 | 352
  Unsatisfactory for Diagnosis | 4 | 2
  Excluded - Slide Preparation Error | 1 | 1

ADVERSE EVENTS:
Arm/Group | SoftPAP | Brush/Spatula
Serious Adverse Events (participants affected / at risk) | 0/348 | 0/355
Other Adverse Events (participants affected / at risk) | 0/348 | 0/355

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No